CLINICAL TRIAL: NCT03519321
Title: Safety and Effectiveness Evaluation of the Minimal Invasive Deformity Correction (MID-C) System in Early Onset Scoliosis
Brief Title: Minimal Invasive Deformity Correction (MID-C) System for Early Onset Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Apifix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF-MID-C-EOS 01-16
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Scoliosis; Scoliosis Idiopathic; Scoliosis;Congenital
Keywords: Early Onset Scoliosis (EOS)
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): MID-C EOS implant will be implanted for the correction of the spine deformity in children found eligible for the study
  Interventions: Device: MID-C

INTERVENTIONS:
Device: MID-C — The MID-C system is being connected to the spine via standard unilateral posterior approach. Pedicle screws above and below the main curve are being used to attach the device to the selected vertebra.

SUMMARY:
Early Onset Scoliosis (EOS) is defined as scoliosis with onset under the age of ten years, regardless of etiology. It is a complex three-dimensional deformity of the spine which can cause significant physical and psychological problems. Currently there are two basic treatment options available for EOS: non-surgical and surgical. ApiFix Ltd. has developed a novel growing rod system for surgical treatment of EOS, the MID-C system. It is indicated for patients with a scoliosis of 35 to 75 degrees Cobb angle

ELIGIBILITY:
Inclusion Criteria:

1. Patients with EOS aged 6-11 years, including idiopathic, syndromic, congenital and low tone neuromuscular diagnoses.
2. Standing x-ray: a single major curve ≤ 8 vertebral segments, 35 to 75 degrees Cobb angle
3. "Normal" or hypokyphotic sagittal contour (T5-T12 ≤ 50⁰ degrees)
4. Primary curve should be reduced to < 35 degrees Cobb angle on lateral bending/traction/stretch x-ray- the residual rigid segment must be ≤ 35 degrees
5. Patients with ≤ 25 degrees trunk rotation based on Scoliometer measurement
6. Subject in good general health
7. Subject and both subject's guardians/legal representatives are willing to sign a written informed consent form

Exclusion Criteria:

1. EOS with more than one structural curve or a single curve involving more than 8 segments
2. High tone neuromuscular diagnoses
3. Primary curve cobb angle > 75 degrees
4. Kyphosis > 50 degrees
5. Previous scoliosis surgery
6. Neural axis abnormality observed by an MRI scan
7. Known allergy to titanium
8. Active systemic disease, such as AIDS, HIV, or active infection
9. Systemic disease that would affect the subject's welfare or overall outcome of the study.
10. Severely mentally compromised

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Maintenance of the major curvature ≤ 50 degrees at 24 months | 24 months
  curve progression will be evaluated by X-ray as in the standard of care

SECONDARY OUTCOMES:
No progression of the primary curve ≥ 10 degrees Cobb angle from correction at time of surgery over time at all follow-up visits | 6 months, 12 months, 24 months
  curve progression will be evaluated by X-ray as in the standard of care
No progression of the secondary (compensatory) curves ≥ 50 degrees Cobb angle over time at all follow-up visits | 6 months, 12 months, 24 months
  curve progression will be evaluated by X-ray as in the standard of care
Blood loss during surgery | Baseline - week 0
  Data will be collected from the hospital surgery records
Duration of surgery | Baseline - week 0
  Data will be collected from the hospital surgery records
Duration of hospitalisation | Baseline - week 0
  Data will be collected from the hospital records
Number of reoperations | 6 Weeks, 3 months, 6 months, 12 months, 24 months
  in case the patient requires a re-operation it will be documented in the study CRF

OTHER OUTCOMES:
Device related serious adverse events | 6 Weeks, 3 months, 6 months, 12 months, 24 months
  AE will be monitored routinely

CONTACTS AND LOCATIONS:
Overall Officials: Ron El-Hawary, MD, Study Director — Chief of Orthopaedics. IWK Health Centre.Associate Professor, Dpt. of Surgery, Dalhousie University, Canada; Ioanna Paspati, MD, Principal Investigator — Spine surgeon
Locations (1):
- Paidon Pentelis Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No